CLINICAL TRIAL: NCT06070532
Title: A Patient Sponsored Ongoing Open-label Single-arm, Safety and Efficacy, Phase I/IIa Clinical Study of Cellcolabs' Human Allogeneic Bone-marrow-derived Mesenchymal Stromal Cell Product (StromaForte) in Patients With Aging Frailty
Brief Title: A Study of Human Allogeneic Bone-marrow-derived Mesenchymal Stromal Cell Product (StromaForte) in Patients With Aging Frailty
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellcolabs Clinical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MROS/220622/INDTP
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): 12 female or male patients suffering from aging frailty
  Interventions: Biological: Human Allogeneic Bone-Marrow-Derived Mesenchymal Stromal Cell Product (StromaForte)

INTERVENTIONS:
Biological: Human Allogeneic Bone-Marrow-Derived Mesenchymal Stromal Cell Product (StromaForte) — 100 x 106 allogeneic bone marrow (BM)-derived Mesenchymal Stromal Cell (MSC) formulated in sodium chloride supplemented with human serum albumin to be given via slow intravenous infusion 100 million cells in approximately 30 min

SUMMARY:
The goal of this phase I/II clinical trial is to evaluate the safety and tolerability of intravenous infusion of human allogeneic bone-marrow-derived mesenchymal stromal cell product StromaForte in patients with aging frailty. The main questions it aims to answer are:

To assess the safety and tolerability after 28 days of injection by reporting the number of adverse events assessed by Common Terminology Criteria For Adverse Events (CTCAE)

Observe the change in inflammatory markers from baseline to 6 months (baseline to 28, 84, and 168 days post-infusion.)

Participants will receive 100 x 106 allogeneic bone marrow (BM)-derived Mesenchymal Stromal Cell (MSC) formulated in sodium chloride supplemented with human serum albumin to be given via slow intravenous infusion 100 million cells in approximately 30 min

DETAILED DESCRIPTION:
Frailty is a geriatric syndrome characterized by weakness, weight loss, and low activity that is associated with adverse health outcomes. One major factor proposed to contribute to frailty and related epigenetic dysregulation is stem cell loss. In order to treat this multifactorial dysregulation, stem cell therapy is an interesting strategy, and MSCs are a particularly tempting candidate. MSCs are an immune-privileged somatic progenitor cell type that is multipotent, self-renewing, and relatively simple to harvest (bone marrow harvest), isolate, and grow. MSCs are proven to regulate the body's immune response in many diseases and exert anti-inflammatory effects. These immunomodulatory properties are mediated via paracrine mechanisms. Following their discovery over 50 years ago, mesenchymal stromal cells (MSCs) have become one of the most studied cellular therapeutic products by both academia and industry due to their regenerative potential and immunomodulatory properties. The promise of MSCs as a therapeutic modality has been demonstrated in a number of preclinical data as well as in clinical setting. StromaForte cells which will be used in this study are developed within CELLCOLABS AB and were generated following the same protocol established over the last 20 years by scientists CELLCOLABS AB at the Karolinska Institute in Sweden. MSCs showed a very promising effect in patients including vocal folds, GVHD, ARDS, multiple sclerosis and recently in patients severely infected with COVID virus The currently completed in vivo studies on rats, rabbits and mice models showed that MSCs could attenuate sarcopenia via increasing skeletal muscle weight and myofiber cross-sectional area. The physical performance including muscle strength aswell as endurance were significantly enhanced. In addition, MSCs have the capability to activate resident skeletal muscle stem cells, which lead to myogenesis and differentiation of muscle tissues. The positive results provide novel insights into sarcopenia intervention, suggesting a potential role for MSC therapy in aging frailty as well as injected doses allogeneic human BM derived MSCs were well tolerated with no treatment-related deaths, biological or neurological changes. No tumor of human origin was detected up to 6 months following administration. These studies demonstrated safety and tolerability of the MSCs. Based on the above results of preclinical studies, it is planned to conduct this study which has been designed to evaluate the safety of intravenous human allogeneic bone marrow-derived mesenchymal stromal cell product StromaForte in frail patients before further clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and comply with all procedures required by the protocol
* Aged > 60 and < 85 years at the time of signing the informed consent form
* Have a Canadian Study on Health and Aging (CSHA) Clinical Frailty Scale score of 5 "mildly frail" or 6 "moderately frail"
* Have a 6-minute walk distance of > 200m and < 400 m
* Have a serum TNF-alpha level >2.5 pg/m

Exclusion Criteria:

1. Unwilling or unable to perform any of the assessments required by the protocol
2. Have a diagnosis of any disabling neurologic disorder, including, but not limited to, Parkinson's disease, Amyotrophic Lateral Sclerosis, multiple sclerosis, cerebrovascular accident with residual deficits (e.g., muscle weakness or gait disorder), or diagnosis of dementia
3. Have a score of 24 or lower on the Mini Mental State Examination (MMSE)
4. Have poorly controlled blood glucose levels (HbA1c >8.0%).
5. Have a clinical history of malignancy within 2.5 years (i.e., patients with prior malignancy must be cancer free for 2.5 years) except curatively treated basal cell carcinoma, melanoma in situ, or cervical carcinoma.
6. Have any condition that limits lifespan to < 1 year according to the Principal Investigator's discretion
7. Have autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus).
8. Undergoes chronic immunosuppressant therapy such as high-dose corticosteroids or TNF-alpha antagonists (prednisone use at doses of < 5 mg daily is allowed)
9. Hepatitis B virus positive
10. Viraemic Hepatitis C virus, HIV-1/2 or syphilis positive
11. Have a resting blood oxygen saturation of <93% (measured by pulse oximetry).
12. Known or suspected alcohol or drug abuse within three years preceding Screening
13. Have a known hypersensitivity to dimethyl sulfoxide (DMSO).
14. An organ transplant recipient (other than transplantation for corneal).
15. Actively listed (or expected future listing) for transplant of any organ (other than corneal transplant).
16. Have any clinically important abnormal screening laboratory values, including, but not limited to: i. Haemoglobin <10.0 g/dL, ii. White blood cell <2,500/ul, or platelet count <100,000/ul iii. Liver dysfunction evidenced by enzymes (AST and ALT) > 3 times the upper limit of normal (ULN)
17. Coagulopathy with an international normalized ratio (INR) >1.3 is not due to a reversible cause (e.g., warfarin and/or Factor Xa inhibitors).
18. Uncontrolled hypertension (resting systolic blood pressure >180 mm Hg or diastolic blood pressure of > 110 mm Hg at screening)
19. Have unstable angina pectoris, uncontrolled or severe peripheral artery disease within the previous 3 months.
20. Have congestive heart failure defined by New York Heart Association (NYHA) Class III or IV, or an ejection fraction of <25%.
21. Have a coronary artery bypass surgery, angioplasty, peripheral vascular disease revascularization, or a myocardial infarction within the previous 3 months
22. Have severe pulmonary dysfunction: acute exacerbation of chronic obstructive lung disease stage III or IV (Gold classification), and/or PaO2 levels <60 mmHg.
23. Have a partial ileal gastric bypass or other significant intestinal malabsorption.
24. Have advanced liver or renal disease
25. Have cognitive or language barriers that prohibit obtaining informed consent or any study elements.
26. Currently hospitalized or living in an assisted living facility or a long-term care facility.
27. Currently participating (or participated within the previous 30 days of consent) in an investigational therapeutic or device trial.
28. Have a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the patient's participation for the full duration of the study

Ages: 60 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of intravenous infusion of human allogeneic bone-marrow-derived mesenchymal stromal cell product Stromaforte | Post 28 day infusion
  To assess the safety and tolerability after 28 days of injection by reporting the number of adverse events assessed by Common Terminology Criteria For Adverse Events (CTCAE) which is the Incidence of any treatment-emergent serious adverse events (TE-SAEs), defined as the composite of death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities determined per the Investigator's judgment

SECONDARY OUTCOMES:
Change in tumor necrosis factor α (TNF-α) | From baseline to 6 months
  Change in tumor necrosis factor α TNF-α from baseline to 6 months (baseline to 28, 84, and 168 days post-infusion.)
Change in C Reactive Protein (CRP) | From baseline to 6 months
  Change in C Reactive Protein (CRP) from baseline to 6 months (baseline to 28, 84, and 168 days post-infusion.
Change in Interleukin-6 (IL-6) | From baseline to 6 months
  Change in Interleukin-6 (IL-6) from baseline to 6 months (baseline to 28, 84, and 168 days post-infusion.
Change in Complete Blood Count (CBC) in peripheral blood with differential | From baseline to 6 months
  Change in Complete Blood Count (CBC) in peripheral blood with differential from baseline to 6 months (baseline to 28, 84, and 168 days post-infusion.

OTHER OUTCOMES:
Change in the 6-minute walk test (6-MWT) | From baseline to 6 months
  Change in the 6-minute walk test (6-MWT) from baseline to 28, 84 and 168 days post infusion
Change in hand grip strength (dynamometry) | From baseline to 6 months
  Change in hand grip strength (dynamometry) from baseline to 84 and 168 days post-infusion
Change in EQ-5D-3L | From baseline to 6 months
  Change in EQ-5D-3L from baseline to 84, and 168 days post-infusion
Change in Multidimensional Fatigue Inventory (MFI) | From baseline to 6 months
  Change in Multidimensional Fatigue Inventory (MFI) from baseline to 84, and 168 days post-infusion
Change in 36-Item Short Form health survey (SF-36) | From baseline to 6 months
  Change in 36-Item Short Form health survey (SF-36) from baseline to 84, and 168 days post-infusion
Change in the Mini Mental State Examination | From baseline to 6 months
  Change in the Mini Mental State Examination (MMSE) criteria after 6 months
Change in cell composition of peripheral blood | From baseline to 6 months
  Change in cell composition of peripheral blood as well as plasma from baseline to 28 days, 84 days, and 168 days post-infusion

CONTACTS AND LOCATIONS:
Locations (1):
- To be decided, Nassau, The Bahamas

IPD SHARING:
Plan to Share IPD: Undecided